CLINICAL TRIAL: NCT01412762
Title: Measuring Patient Expectations for Thyroid Surgery: Development of a Patient-Reported Outcomes Instrument
Brief Title: Measuring Patient Expectations for Thyroid Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-087
Record Dates: First submitted 2011-08-03; First posted 2011-08-09 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Cancer
Keywords: Surgery; interview; 11-087
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patient interviews: We aim to interview 15 patients with confirmed thyroid malignancy both pre- and postoperatively, for a total of 30 interviews. For the expansion of this study, we will accrue 25 patients with biopsy-proven thyroid cancer undergoing thyroidectomy to be educated with the CITSAV application prior to surgery.
  Interventions: Behavioral: patient interviews; Behavioral: CITSAV survey

INTERVENTIONS:
Behavioral: patient interviews — The pre-operative interview will be within 4 weeks of planned surgery and the postoperative interview within 8 weeks of surgery completion. This initial study is designed to develop an instrument to measure patient preoperative expectations in this patient population.
Behavioral: CITSAV survey — Individual semi-structured qualitative interviews will be conducted with a total of 10 patients and 5 clinicians during this phase to identify and discuss levels of satisfaction, level of burden, potential obstacles to implementation, as well as suggestions for improving the intervention

SUMMARY:
The purpose of this study is to learn more about what patients undergoing surgery for thyroid cancer expect from their surgery. Your input may help us to better prepare and inform patients about their disease and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* English speaking
* Patients with confirmed thyroid malignancy confirmed by preoperative fine needle biopsy (any stage) planned for surgical excision

Exclusion Criteria:

* Inability to speak or understand English
* Inability to provide meaningful informed consent due to physical, cognitive, or psychiatric disability
* Prior thyroid surgery
* Prior radioactive iodine treatment, external beam radiation or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for thyroid cancer will be recruited by the attending Head and Neck Surgeons and Research Study Assistants in the Head and Neck Clinic
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To establish a patient-reported outcomes tool for measuring preoperative expectations in patients undergoing surgery for thyroid cancer. | 2 year
  This will be done by conducting qualitative semistructured interviews with 15 thyroid cancer patients (pre- and postoperatively) to identify recurring themes about their expectations regarding thyroid surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Patel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm